CLINICAL TRIAL: NCT01848093
Title: Molekularbiologische Eigenschaften Des Sputums während Einer Pulmonalen COPD Exacerbation
Brief Title: Mucin Concentration in Sputum From COPD Patients During a Pulmonary Exacerbation
Acronym: mucinCOPDex
Status: Withdrawn | Type: Observational
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Other Study IDs: 160/08
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2013-05

CONDITIONS: COPD
Keywords: lung; airway; pulmonary exacerbation; mucus
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD exacerbation: COPD Stadium 2 and 3 during pulmonary exacerbation
  sputum collection
  Interventions: Other: sputum collection

INTERVENTIONS:
Other: sputum collection — collecting of spontaneous sputum from the patient

SUMMARY:
chronic obstructive pulmonary disease (COPD) is typically associated with mucus hypersecretion in the airways. In health, mucin is the major macromolecular component and is responsible for the protective and clearance properties of the mucus gel. In a recent study the investigators found that mucins are decreased and unstable in the sputum of adult cystic fibrosis (CF) patients.

In this study the investigators want to investigate the differences on the mucin quantity and quality of airway secretions during pulmonary exacerbation of patients with COPD.

DETAILED DESCRIPTION:
We hypothesize that during an exacerbation the mucin amount is increasing.

The aim of this study is to evaluate the molecular (mucins) and structure properties (mucin-stability) of the airway secretions in COPD related to the severity of the disease.

We characterize sputum composition of patients with pulmonary exacerbations. Using gel electrophoresis, with specific antibodies we will analyze MUC5AC and MUC5B mucins.

The significance of these studies is that they will give us novel information about the pathogenesis of chronic inflammatory airway diseases, provide tools for assessing the progression of lung disease, and most critically, will identify novel opportunities and targets for therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* forced expiratory volume at one second (FEV1) < 80%
* sputum production
* clinical likely hood of exacerbation

Exclusion Criteria:

* FEV1 > 80% or < 30%
* increased systemic inflammation
* susceptibility of pneumonia
* need for antibiotic treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients Stadium 2-3 during pulmonary exacerbation
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
mucin concentration | 2 month
  analyzing mucin concentration by western

SECONDARY OUTCOMES:
mucin stability | 2 month
  analyzing mucin stability at 37C over 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Markus Henke, MD, Principal Investigator — University Marburg
Locations (2):
- Germany (2):
  - pulmonary department, University Marburg, Marburg
  - University Marburg, Marburg

REFERENCES:
- [Background] Henke MO, Renner A, Huber RM, Seeds MC, Rubin BK. MUC5AC and MUC5B Mucins Are Decreased in Cystic Fibrosis Airway Secretions. Am J Respir Cell Mol Biol. 2004 Jul;31(1):86-91. doi: 10.1165/rcmb.2003-0345OC. Epub 2004 Feb 26. PMID 14988081
- [Background] Henke MO, John G, Rheineck C, Chillappagari S, Naehrlich L, Rubin BK. Serine proteases degrade airway mucins in cystic fibrosis. Infect Immun. 2011 Aug;79(8):3438-44. doi: 10.1128/IAI.01252-10. Epub 2011 Jun 6. PMID 21646446
- [Background] Henke MO, John G, Germann M, Lindemann H, Rubin BK. MUC5AC and MUC5B mucins increase in cystic fibrosis airway secretions during pulmonary exacerbation. Am J Respir Crit Care Med. 2007 Apr 15;175(8):816-21. doi: 10.1164/rccm.200607-1011OC. Epub 2007 Jan 25. PMID 17255563